CLINICAL TRIAL: NCT03950206
Title: Intraoperative Assessment of Ureteral Perfusion Using Indocyanine Green Angiography in Women Submitted to Laparoscopic Surgery for Endometriosis
Brief Title: Intraoperative Assessment of Ureteral Perfusion in Women With Endometriosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to terminate the trial
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Renato Seracchioli, Principal Investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICG and endometriosis
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2019-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Ureters; Indocyanine green angiography
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with endometriosis (Other): Women undergoing laparoscopic surgery for endometriosis
  Interventions: Other: Indocyanine green angiography

INTERVENTIONS:
Other: Indocyanine green angiography — Intravenous ICG (PULSION Medical Systems SE, Feldkirchen, Germany) will be used for the intraoperative evaluation of ureteral vascularization. Twenty-five milligrams of indocyanine green will be diluted in 10 ml of soluble water, and a bolus of 0.25 mg/Kg will be injected through a peripheral vein. During laparoscopy, a NIR camera-head (KARL STORZ Gesellschaft Mit Beschränkter Haftung& Co., Tuttlingen, Germany) will be used to visualize the ureteral vascularization.

SUMMARY:
Deep infiltrating endometriosis (DIE) is a severe form of endometriosis in which lesions affect retroperitoneal tissue and pelvic organs wall. It is often characterized by pain (dysmenorrhea, dysuria, dyspnea, dyspareunia, and chronic pelvic pain) and infertility, drastically impacting on women' quality of life. It is typically multifocal, involving uterosacral ligaments, the upper third of posterior vaginal wall, bowel, bladder, and ureters.

Indocyanine green (ICG) is an anionic tricarbocyanine molecule able to bind to plasma proteins into the vascular system and to become fluorescent if excited by near-infrared light (NIR). NIR-ICG imaging is used in gynecology for the intraoperative diagnosis of occult peritoneal and deep endometriosis at white light and to assess tissue perfusion and guide surgical strategy.

DETAILED DESCRIPTION:
Patients with clinical and trans-vaginal / abdominal ultrasound diagnosis of deep endometriosis, undergoing surgery for the removal of endometriotic lesions are included in the study.

Ureter perfusion will be intraoperatively assessed using indocyanine green angiography.

After surgery, patients will be included in the post-operative follow-up, as usual in our clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic surgery for endometriosis
* informed consent to participate in the study

Exclusion Criteria:

* known or suspected allergy to iodide
* history of active pelvic infection
* presence of intra-abdominal or pelvic malignancy
* pelvic radiation therapy
* hyperthyroidism
* liver dysfunction
* serum creatinine > 2.0 mg/dL

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety: Clavien-Dindo Classification (from Grade I to V) | From the surgery time, assessed up to 7 days after surgery
  Evaluation of feasibility and safety of indocyanine green angiography in women submitted to laparoscopic surgery for endometriosis, considering complications using Clavien-Dindo Classification (from Grade I to V)

SECONDARY OUTCOMES:
Ureteral vascularization | Intraoperative
  Evaluation of ureteral vascularization using indocyanine green angiography in women submitted to laparoscopic surgery for endometriosis

CONTACTS AND LOCATIONS:
Locations (1):
- Diego Raimondo, Bologna, BO, Italy

REFERENCES:
- [Derived] Raimondo D, Borghese G, Mabrouk M, Arena A, Ambrosio M, Del Forno S, Degli Esposti E, Casadio P, Mattioli G, Mastronardi M, Seracchioli R. Use of Indocyanine Green for Intraoperative Perfusion Assessment in Women with Ureteral Endometriosis: A Preliminary Study. J Minim Invasive Gynecol. 2021 Jan;28(1):42-49. doi: 10.1016/j.jmig.2020.04.004. Epub 2020 Apr 10. PMID 32283326